CLINICAL TRIAL: NCT07390721
Title: Effects of Diaphragmatic Kinesio Taping-Assisted HIIT Exercises on Aerobic Capacity, Anaerobic Capacity, and Balance in Trained Individuals
Brief Title: Diaphragmatic Kinesio Taping With HIIT in Trained Individuals
Acronym: DKT-HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Collaborators: Health Institutes of Turkey (Other Government); Uludag University (Other)
Responsible Party: Principal Investigator, Dursun Alper YILMAZ, Res. Asst., Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BUU-FIZ-HIIT-KT-2025
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Postural Balance; Physical Fitness; Healthy Volunteers
Keywords: VO2max; Balance; Kinesio Taping; High-Intensity Interval Training; Anaerobic Performance
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a HIIT plus diaphragmatic kinesio taping group or a HIIT-only control group, and both groups are followed in parallel for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT + Diaphragmatic Kinesio Taping (Experimental): Participants perform an 8-week HIIT program and receive diaphragmatic kinesio taping before each training session.
  Interventions: Behavioral: High-Intensity Interval Training (HIIT); Other: Diaphragmatic Kinesio Taping
- HIIT Only (Active Comparator): Participants perform the same 8-week HIIT program without kinesio taping.
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: High-Intensity Interval Training (HIIT) — Participants perform an 8-week supervised high-intensity interval training program on a cycle ergometer, three times per week. Each session includes warm-up, alternating high- and low-intensity intervals targeting 85-95% of maximal heart rate, and cool-down.
Other: Diaphragmatic Kinesio Taping — Elastic kinesio tape is applied to the diaphragmatic region before each training session using a standardized technique to support inspiratory muscle activity and facilitate breathing.
  Arms: HIIT + Diaphragmatic Kinesio Taping

SUMMARY:
This study examines whether adding diaphragmatic kinesio taping to high-intensity interval training (HIIT) improves physical performance in trained individuals. Participants will be randomly assigned to one of two groups. One group will perform an 8-week HIIT program on a cycle ergometer. The other group will follow the same HIIT program and will also receive diaphragmatic kinesio taping before each exercise session. The taping is applied to support breathing muscles and may help improve oxygen use during exercise.

Before and after the training period, participants will undergo tests to measure aerobic capacity (VO₂max), anaerobic power (Wingate test), balance (Y-Balance test), lung function (spirometry), body composition, and heart rate responses. The results of this study will help determine whether diaphragmatic kinesio taping provides additional benefits when combined with HIIT training.

DETAILED DESCRIPTION:
This randomized controlled experimental study evaluates the combined effects of high-intensity interval training (HIIT) and diaphragmatic kinesio taping on aerobic capacity, anaerobic performance, balance, and respiratory function in trained adults.

HIIT is known to elicit strong cardiovascular, metabolic, and neuromuscular adaptations through repeated short bouts of high-intensity exercise interspersed with recovery periods. Although HIIT is widely used to improve aerobic and anaerobic fitness, the potential contribution of respiratory muscle support strategies to enhance these adaptations remains largely unexplored. Diaphragmatic kinesio taping is a non-invasive method that may facilitate inspiratory muscle activation, improve breathing mechanics, and support oxygen utilization during exercise.

The main objective of this study is to determine whether adding diaphragmatic kinesio taping to a structured HIIT program produces superior improvements in aerobic capacity, anaerobic power, balance, and pulmonary function compared with HIIT alone. The study also aims to explore whether this combined approach influences post-exercise balance and neuromuscular control, which are relevant for both performance and injury prevention.

Participants aged 18-35 years with at least six months of regular training experience will be randomly assigned to either an experimental group (HIIT with diaphragmatic kinesio taping) or a control group (HIIT only). Both groups will complete an eight-week training program consisting of three supervised sessions per week on a cycle ergometer. Exercise intensity will be individually prescribed to reach 85-95% of maximal heart rate during high-intensity intervals, with active recovery periods at lower intensities.

In the experimental group, diaphragmatic kinesio taping will be applied before each training session using a standardized technique designed to support the primary respiratory muscles. The control group will follow the same HIIT protocol without taping. No changes to participants' usual training outside the study will be encouraged.

Assessments will be performed before and after the intervention under standardized laboratory conditions. Aerobic capacity will be estimated using a ramp test protocol, anaerobic performance will be evaluated using a short maximal cycling test, and balance will be assessed through validated static and dynamic balance tests. Pulmonary function, body composition, and heart rate responses will also be recorded to provide a comprehensive evaluation of physiological adaptations.

The study is conducted at Bursa Uludag University Faculty of Medicine, Department of Physiology, and has received approval from the institutional ethics committee. All participants will provide written informed consent prior to participation. The findings of this study are expected to contribute to evidence-based exercise programming by clarifying whether respiratory muscle support through diaphragmatic kinesio taping enhances the benefits of HIIT in trained individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* Male or female trained individuals
* At least 6 months of regular training history
* Training at least 3-5 days per week
* Estimated VO₂max ≥ 50 ml/kg/min
* No known contraindication to high-intensity exercise
* No allergy or skin condition preventing kinesio taping
* Able to provide written informed consent

Exclusion Criteria:

* History of cardiovascular, respiratory, or metabolic disease (e.g., asthma, COPD, diabetes, heart disease)
* Major musculoskeletal injury or surgery within the past 6 months
* Any pathology affecting diaphragm or respiratory muscles
* Active smoking or substance abuse
* Use of performance-enhancing drugs
* Skin disease in the abdominal region

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Aerobic Capacity (VO₂max) | From baseline to the end of the 8-week intervention
  Change in maximal oxygen uptake estimated from a ramp exercise test performed on a cycle ergometer at baseline and after the 8-week intervention.
Anaerobic Performance (Wingate Test) | Baseline and after 8 weeks
  Change in peak power, mean power, and fatigue index measured by the 30-second Wingate anaerobic test at baseline and after the 8-week intervention.
Dynamic Balance (Y-Balance Test) | Baseline and after 8 weeks
  Change in normalized reach distances in the anterior, posteromedial, and posterolateral directions measured by the Y-Balance Test at baseline and after the 8-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fadıl Özyener, Prof. Dr., Study Director — Uludag University
Locations (1):
- Bursa Uludag University, Bursa, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly because the dataset contains potentially identifiable information and participants did not provide consent for open data sharing. Aggregated and anonymized results will be made available through publications.

REFERENCES:
- [Result] Seiler S. It's about the long game, not epic workouts: unpacking HIIT for endurance athletes. Appl Physiol Nutr Metab. 2024 Nov 1;49(11):1585-1599. doi: 10.1139/apnm-2024-0012. Epub 2024 Jul 30. PMID 39079169
- [Result] Schvambach M, Isoppo KDS. Immediate effects of Kinesio Taping (R) on respiratory parameters in healthy individuals. J Bodyw Mov Ther. 2024 Oct;40:1153-1157. doi: 10.1016/j.jbmt.2024.07.030. Epub 2024 Jul 11. PMID 39593427
- [Result] Guo Z, Li M, Cai J, Gong W, Liu Y, Liu Z. Effect of High-Intensity Interval Training vs. Moderate-Intensity Continuous Training on Fat Loss and Cardiorespiratory Fitness in the Young and Middle-Aged a Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2023 Mar 8;20(6):4741. doi: 10.3390/ijerph20064741. PMID 36981649
- [Result] Ito S. High-intensity interval training for health benefits and care of cardiac diseases - The key to an efficient exercise protocol. World J Cardiol. 2019 Jul 26;11(7):171-188. doi: 10.4330/wjc.v11.i7.171. PMID 31565193
- [Result] Wang X, Soh KG, Samsudin S, Li L, Liu C, Sun M, Ma S. Effects of high-intensity training on jumping performance among athletes: a systematic review with meta-analysis. Sci Rep. 2025 Jan 13;15(1):1763. doi: 10.1038/s41598-024-83161-5. PMID 39800767
- [Result] Seo Y, Lee Y, Son S, Lee J, Park J, Lee D, Seon SY, Yun S. Does Kinesio Taping Enhance Exercise Performance and Recovery in Healthy Males Under Heat Stress? J Clin Med. 2025 Apr 11;14(8):2631. doi: 10.3390/jcm14082631. PMID 40283460